CLINICAL TRIAL: NCT06919939
Title: Phase 2 Study of Epcoritamab in Combination With Loncastuximab Tesirine in Relapsed/Refractory Large B-cell Lymphoma
Brief Title: Epcoritamab in Combination With Loncastuximab Tesirine in Relapsed/Refractory Large B-cell Lymphoma
Acronym: EPCOR+LONCA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: ADC Therapeutics S.A. (Industry); Genmab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20241140
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Large B-cell Lymphoma; Relapse
MeSH Terms: conditions — Recurrence | interventions — loncastuximab tesirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EPCOR in combination with LONCA Treatment Group (Experimental): Participants in the Epcoritamab (EPCOR) in combination with Loncastuximab (LONCA) treatment group will receive up to 4 cycles of combination EPCOR and LONCA therapy, and an additional 8 cycles of EPCOR therapy, for a total of twelve treatment cycles. Cycles 1 through 3 last 21 days each; cycles four through 12 last 28 days each. Protocol therapy will last approximately 12 months.
  Total participation duration is approximately 3 years.
  Interventions: Drug: Epcoritamab; Drug: Loncastuximab Tesirine

INTERVENTIONS:
Drug: Epcoritamab — Epcoritamab will be administered via subcutaneous injection at the following dose levels and schedule over a total of twelve cycles:
  * Cycle 1 Day 1: Step-up dose of 0.16 mg
  * Cycle 1 Day 8: Step-up dose of 0.80 mg
  * Cycle 1 Day 15: First full dose of 48 mg.
  * Cycles 2 through 4 Days 1, 8 and 15: 48 mg
  * Cycles 5 through 12 Days 1 and 15: 48 mg
  Other Names: Epkinly
Drug: Loncastuximab Tesirine — Loncastuximab will be administered intravenously (IV) at the following dose level and schedule over a total of four cycles:
  * Cycles 1 and 2 Day 1: 120 mcg/kg
  * Cycles 3 and 4 Day 1: 75 mcg/kg
  * Cycle 4 Day 22: 75 mcg/kg
  Other Names: Loncatuximab; Zynlonta

SUMMARY:
The purpose of this study is to determine whether combining Loncastuximab Tesirine with Epcoritamab is tolerable and effective for reducing and/or eliminating lymphoma cells in the body.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 years or older at the time of signing informed consent.
2. Able and willing to sign the informed consent form (ICF).
3. Ability to comply with the trial protocol.
4. Relapsed/refractory (r/r) large B-cell lymphoma (LBCL) as determined by the local hematopathology laboratory from the following diagnoses by 2016 World Health Organization (WHO) classification of lymphoid neoplasms (Swerdlow et al., 2016):

   1. LBCL or DLBCL, not otherwise specified (NOS)
   2. High-grade B-cell lymphoma (NOS or double/triple hit [technically classified in WHO 2016 as high-grade B-cell lymphoma (HGBCL), with Myc and B-cell lymphoma 2 (BCL2) and/or B-cell lymphoma 6 (BCL6) translocations])
   3. Transformed from follicular lymphoma, marginal zone lymphoma (MZL), and nodular lymphocyte predominant Hodgkin lymphoma
   4. Follicular lymphoma stage 3B
   5. Primary mediastinal B-cell lymphoma previously treated with checkpoint inhibitor Note: Relapsed disease is defined as disease that has recurred ≥6 months after completion of therapy. Refractory disease is defined as disease that either progressed during therapy or progressed within 6 months (<6 months) of completion of therapy.
5. Participants who have received at least one prior systemic therapy for LBCL including anti-cluster of differentiation 20 (anti-CD20) monoclonal antibody and anthracycline-containing therapy.
6. Measurable disease by 2014 Lugano Classification. (Participants who have measurable disease, defined as at least 1 bi-dimensionally measurable nodal lesion, defined as >1.5 cm in its longest dimension, or at least 1 bi-dimensionally measurable extra nodal lesion, defined as >1.0 cm in its longest dimension.)
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 to 2.
8. Adequate hematologic, hepatic, and renal function tested within 6 weeks prior to the start of therapy (values must not be achieved with growth factors within 72 hs):

   1. Absolute neutrophil count (ANC) ≥ 1.0 × 10^9 cells/L
   2. Hemoglobin ≥8.0 g/dL without blood transfusion in the past week
   3. Platelet count ≥75 × 10^9 platelets/L or ≥ 50 × 10^9 platelets/L if bone marrow involvement or splenomegaly
   4. Total bilirubin ≤1.5 × upper limit normal (ULN). Participants with documented history of Gilbert's syndrome and in whom total bilirubin elevations are accompanied by elevated indirect bilirubin are eligible (≤3x institutional ULN if lymphoma involvement of the liver).
   5. Alanine transaminase (ALT)/aspartate aminotransferase (AST) ≤3.0 × ULN or ≤5 × ULN in the presence of liver involvement by lymphoma.

      * i. Creatinine within normal institutional limits, or calculated creatinine clearance ≥40 mL/min by the Cockcroft-Gault Equation or other institutional standard methods
9. Willingness to avoid pregnancy during the trial and for at least 12 months after the last dose of the trial intervention.
10. Patients with history of human immunodeficiency virus (HIV) are eligible, provided they are stable on anti-retroviral therapy, have cluster of differentiation 4 (CD4) count ≥200/µL, and have an undetectable viral load. Note: HIV test is optional.
11. Life expectancy of at least 12 weeks
12. For patients receiving glucocorticoid treatment at screening: treatment must be tapered down and administered with a maximum of 25 mg daily in the last 14 days before the first dose of epcoritamab.

Exclusion Criteria:

1. Primary central nervous system (CNS) lymphoma or known CNS involvement by lymphoma at screening as confirmed by magnetic resonance imaging (MRI)/computed tomography (CT) scan (brain) and, if clinically indicated, by lumbar puncture.
2. Prior treatment with anti-cluster of differentiation 19 (anti-CD19) chimeric antigen receptor T-cell (CAR-T) therapy
3. Prior exposure to bispecific T-cell engaging antiCD20XCD3 antibodies
4. Prior autologous or allogenic stem cell transplant
5. Known clinically significant pulmonary disease, including:

   1. Pulmonary fibrosis affecting patient's exercise tolerance.
   2. Chronic obstructive pulmonary disease (COPD) affecting patient's exercise tolerance.
6. Known clinically significant cardiac disease, including:

   1. Onset of unstable angina pectoris within 6 months of signing ICF
   2. Acute myocardial infarction within 6 months of signing ICF
   3. Congestive heart failure (grade III or IV as classified by the New York Heart Association
7. Pregnant or breast feeding
8. Inadequate recovery from toxicity and/or complications from a major surgery before starting therapy.
9. Chronic or current active infectious disease (including severe acute respiratory syndrome (SARS) coronavirus 2 (CoV-2) requiring systemic antibiotics, antifungal, or antiviral treatment or any major episode of infection requiring treatment with intravenous (IV) antibiotics within 2 weeks of Day 1 of Cycle 1.
10. Exposure to a live vaccine within 30 days of administration or anticipation that a live attenuated vaccine will be required during the study.

    1. Inactivated influenza vaccinations may be given during the influenza season.
    2. An approved coronavirus disease 2019 (COVID-19) vaccine (messenger ribonucleic acid (mRNA), inactivated virus, and replication deficient viral vector vaccines) is allowed.
11. Active hepatitis B infection

    a. Patients who are hepatitis B surface antigen (HbsAg) negative and hepatitis B core antibody (HbcAb) positive must be negative for hepatitis B virus (HBV) polymerase chain reaction (PCR) to be eligible for study participation
12. Active hepatitis C infection

    a. Patients who are positive for hepatitis C virus (HCV) antibody must be negative for HCV by PCR to be eligible for study participation
13. Patient has no known active SARS-CoV-2 infection. If a subject has signs/symptoms suggestive of SARS-CoV-2 infection, the patient must have a negative molecular (eg, PCR) test or 2 negative antigen test results at least 24 hours apart.

    Note: SARS-CoV-2 diagnostic tests should be applied following local requirements/recommendations. Patients who do not meet SARS-CoV-2 infection eligibility criteria must be screen-failed and may only rescreen if the following have been met:
    * At least 10 days since first positive test result have passed in asymptomatic patients or at least 10 days since recovery, defined as resolution of fever without use of antipyretics and improvement in symptoms.
14. Patients with severe chronic pulmonary disease, or other serious medical condition which is likely to significantly impair the patient's ability to tolerate the study treatment.
15. Patients with seizure disorder requiring therapy with a last convulsion within two years from enrollment.
16. Patients with impaired decision-making capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2031-02-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Cytokine Release Syndrome (CRS)-related Toxicity after Epcoritamab Administration | Up to 14 months
  The number of participants experiencing Cytokine Release Syndrome (CRS) toxicity associated with Epcoritamab therapy will be reported, including Grades 2, 3 and 4. CRS-related toxicity will be assessed according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria.
Number of Participants Experiencing Immune Effector Cell Associated Neurotoxicity Syndrome (ICANS)-related Toxicity | Up to 14 months
  The number of participants experiencing Immune Effector Cell Associated Neurotoxicity Syndrome (ICANS)-related toxicity including Grades 2, 3 and 4. ICANS-related toxicity will be assessed according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria.
Number of Participants Experiencing Neurologic Toxicities Associated with Epcoritamab | Up to 14 months
  The number of participants experiencing neurologic toxicities associated with Epcoritamab therapy will be reported, including Grades 2, 3 and 4. Neurologic toxicities will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, per physician discretion.
Number of Participants Experiencing Fluid Accumulation Associated with Loncastuximab | Up to 31 weeks
  The number of participants experiencing fluid accumulation associated with Loncastuximab therapy will be reported, including Grades 2, 3 and 4. Fluid accumulation toxicities will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, per physician discretion.
Number of Participants Experiencing Hepatotoxicity Associated with Loncastuximab | Up to 31 weeks
  The number of participants experiencing hepatotoxicity (liver-related toxicity) associated with Loncastuximab therapy including Grades 2, 3 and 4 toxicity. Hepatotoxicity will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, per physician discretion.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 36 months
  Overall response rate is defined as the number of participants with complete metabolic response (CMR) or partial metabolic response (PMR) as the best response. Response will be assessed according to Lugano 2014 criteria.
Partial Metabolic Response (PMR) Rate | Up to 36 months
  PMR rate is defined as the number of participants with partial metabolic response (PMR) as the best response according to Lugano 2014 criteria.
Progression-Free Survival (PFS) | Up to 36 months
  PFS is defined as the elapsed time in months from the start of treatment until disease progression or death, whichever is earlier. Participants who remain alive without progression will be censored at the last documented disease assessment date. Response will assessed according to Lugano 2014 criteria.
Overall Survival (OS) | Up to 36 months
  OS is defined as the elapsed time in months from the start of treatment until death from any cause. Alive participants will be censored at the last date known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Alderuccio, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No